CLINICAL TRIAL: NCT02284464
Title: Steroid Withdrawal and Novo Donor-specific Anti-HLA Antibodies in Renal Transplant Patients: a Prospective, Randomized and Controlled Study in Parallel Groups
Brief Title: Steroid Withdrawal and Donor-specific Anti-HLA Antibodies in Renal Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: Sociedad Andaluza de Trasplantes de Organos y Tejidos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVITAESTEROIDE-12
Record Dates: First submitted 2014-10-16; First posted 2014-11-06 (Estimated); Results first posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2019-12

CONDITIONS: Other Complication of Kidney Transplant; Renal Transplant Rejection
Keywords: Kidney transplant; Immunosuppression; Steroid withdrawal; Donor specific antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Steroids, tacrolimus and mycophenolate (Active Comparator): Normal treatment arm
  Interventions: Drug: Prednisone continuation
- Tacrolimus and mycophenolate (Experimental): Normal treatment for first 90 days, then steroid withdrawal carrying on with the other drugs
  Interventions: Drug: Prednisone withdrawal

INTERVENTIONS:
Drug: Prednisone withdrawal — Withdrawal of steroids
  Arms: Tacrolimus and mycophenolate
Drug: Prednisone continuation — Continuation of steroids
  Arms: Steroids, tacrolimus and mycophenolate

SUMMARY:
Steroids are one of the pillars of immunosuppression for kidney transplant patients but their use is associated with a high rate of complications. Withdrawal of steroids reduces some metabolic and cardiovascular complications, but it may increase the risk of acute rejection. However, little is known about whether steroid withdrawal is associated with the generation of anti-HLA donor-specific antibodies (DSA) and the relation between DSA and clinical and histological data. The aim of this study is to compare the incidence of de novo anti-HLA DSA in stable kidney transplant patients after withdrawing the steroids 3 months after the transplantation as compared with patients who continue with steroids. The hypothesis is that steroid withdrawal will increase the presence of de novo anti-HLA DSA in stable kidney transplant patients

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged over 18 years with no immunological risk (PRA <25% and no DSA) who are receiving their first cadaveric or living kidney transplant.
2. Patients who, three months after the transplantation, are receiving tacrolimus in combination with mycophenolic acid (MPA) or mycophenolate mofetil (MMF) plus steroids, with stable plasma levels of tacrolimus.
3. No clinical or histological immunological dysfunction before randomization
4. No de novo anti-HLA DSA at the time of randomization.
5. Patients who wish to and are able to give written informed consent to participate in the study.
6. For women, agreeing to use efficient contraception during the study.

Exclusion Criteria:

1. Patients who receive a multiorgan transplant.
2. Retransplants.
3. Presence of DSA before the transplant or at the time of randomization.
4. Cold ischemia time >30 hours
5. Patients with serum creatinine >2 mg/dL or proteinuria >1g/day at the time of randomization
6. Prior episode of severe rejection (II-B-III in the Banff/13 classification) prior to randomization.
7. Presence of subclinical rejection on the protocol biopsy prior to randomization
8. Patients with BK-polyomavirus nephropathy at the time of randomization.
9. Patients with recurrent or de novo glomerulonephritis.
10. Patients who are being treated with immunosuppressive drugs other than those in the randomized clinical trial in question.
11. Patients who are positive for the human immunodeficiency virus (HIV) or those who have a severe systemic infection that, in the investigator's judgment, will require continued treatment.
12. Patients with any present or prior (during the previous 5 years) malignant disease, except basal or squamous cell carcinoma that has been excised.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2015-02; Primary Completion 2019-07 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Domingo Hernandez, PhD, Principal Investigator — Carlos Haya Hospital
Locations (5):
- Spain (5):
  - Vall d Hebron Hospital, Barcelona
  - Bellvitge Hospital, Barcelona
  - Carlos Haya Hospital, Málaga
  - Canarias University Hospital, Santa Cruz de Tenerife
  - Dr. Peset Hospital, Valencia

REFERENCES:
- [Background] Miller LW. Cardiovascular toxicities of immunosuppressive agents. Am J Transplant. 2002 Oct;2(9):807-18. doi: 10.1034/j.1600-6143.2002.20902.x. PMID 12392286
- [Background] Marcen R. Immunosuppressive drugs in kidney transplantation: impact on patient survival, and incidence of cardiovascular disease, malignancy and infection. Drugs. 2009 Nov 12;69(16):2227-43. doi: 10.2165/11319260-000000000-00000. PMID 19852526
- [Background] Vincenti F, Schena FP, Paraskevas S, Hauser IA, Walker RG, Grinyo J; FREEDOM Study Group. A randomized, multicenter study of steroid avoidance, early steroid withdrawal or standard steroid therapy in kidney transplant recipients. Am J Transplant. 2008 Feb;8(2):307-16. doi: 10.1111/j.1600-6143.2007.02057.x. PMID 18211506
- [Background] Arnol M, de Mattos AM, Chung JS, Prather JC, Mittalhenkle A, Norman DJ. Late steroid withdrawal and cardiovascular events in kidney transplant recipients. Transplantation. 2008 Dec 27;86(12):1844-8. doi: 10.1097/TP.0b013e31818ffec0. PMID 19104432
- [Background] Opelz G, Dohler B. Association between steroid dosage and death with a functioning graft after kidney transplantation. Am J Transplant. 2013 Aug;13(8):2096-105. doi: 10.1111/ajt.12313. Epub 2013 Jun 10. PMID 23750878
- [Background] Opelz G, Dohler B, Laux G; Collaborative Transplant Study. Long-term prospective study of steroid withdrawal in kidney and heart transplant recipients. Am J Transplant. 2005 Apr;5(4 Pt 1):720-8. doi: 10.1111/j.1600-6143.2004.00765.x. PMID 15760395
- [Background] Gonzalez-Molina M, Gentil MA, Burgos D, Cabello M, Cobelo C, Bustamante J, Errasti P, Franco A, Hernandez D. Effect of long-term steroid withdrawal in renal transplant recipients: a retrospective cohort study. NDT Plus. 2010 Jun;3(Suppl_2):ii32-ii36. doi: 10.1093/ndtplus/sfq064. PMID 20508858
- [Background] Kasiske BL, Chakkera HA, Louis TA, Ma JZ. A meta-analysis of immunosuppression withdrawal trials in renal transplantation. J Am Soc Nephrol. 2000 Oct;11(10):1910-1917. doi: 10.1681/ASN.V11101910. PMID 11004223
- [Background] Pascual J, Quereda C, Zamora J, Hernandez D; Spanish Group for Evidence-Based Medicine in Renal Transplantation. Steroid withdrawal in renal transplant patients on triple therapy with a calcineurin inhibitor and mycophenolate mofetil: a meta-analysis of randomized, controlled trials. Transplantation. 2004 Nov 27;78(10):1548-56. doi: 10.1097/01.tp.0000140969.43761.1f. PMID 15599321
- [Background] Woodle ES, First MR, Pirsch J, Shihab F, Gaber AO, Van Veldhuisen P; Astellas Corticosteroid Withdrawal Study Group. A prospective, randomized, double-blind, placebo-controlled multicenter trial comparing early (7 day) corticosteroid cessation versus long-term, low-dose corticosteroid therapy. Ann Surg. 2008 Oct;248(4):564-77. doi: 10.1097/SLA.0b013e318187d1da. PMID 18936569
- [Background] Terasaki PI, Ozawa M. Predicting kidney graft failure by HLA antibodies: a prospective trial. Am J Transplant. 2004 Mar;4(3):438-43. doi: 10.1111/j.1600-6143.2004.00360.x. PMID 14961999
- [Background] Wiebe C, Gibson IW, Blydt-Hansen TD, Karpinski M, Ho J, Storsley LJ, Goldberg A, Birk PE, Rush DN, Nickerson PW. Evolution and clinical pathologic correlations of de novo donor-specific HLA antibody post kidney transplant. Am J Transplant. 2012 May;12(5):1157-67. doi: 10.1111/j.1600-6143.2012.04013.x. Epub 2012 Mar 19. PMID 22429309
- [Background] Gill JS, Landsberg D, Johnston O, Shapiro RJ, Magil AB, Wu V, Tinckam K, Keown P. Screening for de novo anti-human leukocyte antigen antibodies in nonsensitized kidney transplant recipients does not predict acute rejection. Transplantation. 2010 Jan 27;89(2):178-84. doi: 10.1097/TP.0b013e3181c3503e. PMID 20098280
- [Background] Cantarovich D, De Amicis S, Akl A, Devys A, Vistoli F, Karam G, Soulillou JP. Posttransplant donor-specific anti-HLA antibodies negatively impact pancreas transplantation outcome. Am J Transplant. 2011 Dec;11(12):2737-46. doi: 10.1111/j.1600-6143.2011.03729.x. Epub 2011 Sep 11. PMID 21906255
- [Background] Hoshino J, Kaneku H, Everly MJ, Greenland S, Terasaki PI. Using donor-specific antibodies to monitor the need for immunosuppression. Transplantation. 2012 Jun 15;93(11):1173-8. doi: 10.1097/TP.0b013e31824f3d7c. PMID 22592887
- [Background] Worthington JE, Martin S, Al-Husseini DM, Dyer PA, Johnson RW. Posttransplantation production of donor HLA-specific antibodies as a predictor of renal transplant outcome. Transplantation. 2003 Apr 15;75(7):1034-40. doi: 10.1097/01.TP.0000055833.65192.3B. PMID 12698094
- [Background] Mao Q, Terasaki PI, Cai J, Briley K, Catrou P, Haisch C, Rebellato L. Extremely high association between appearance of HLA antibodies and failure of kidney grafts in a five-year longitudinal study. Am J Transplant. 2007 Apr;7(4):864-71. doi: 10.1111/j.1600-6143.2006.01711.x. PMID 17391129
- [Background] Moreso F, Ibernon M, Goma M, Carrera M, Fulladosa X, Hueso M, Gil-Vernet S, Cruzado JM, Torras J, Grinyo JM, Seron D. Subclinical rejection associated with chronic allograft nephropathy in protocol biopsies as a risk factor for late graft loss. Am J Transplant. 2006 Apr;6(4):747-52. doi: 10.1111/j.1600-6143.2005.01230.x. PMID 16539631
- [Background] Anil Kumar MS, Irfan Saeed M, Ranganna K, Malat G, Sustento-Reodica N, Kumar AM, Meyers WC. Comparison of four different immunosuppression protocols without long-term steroid therapy in kidney recipients monitored by surveillance biopsy: five-year outcomes. Transpl Immunol. 2008 Nov;20(1-2):32-42. doi: 10.1016/j.trim.2008.08.005. Epub 2008 Sep 4. PMID 18773960
- [Derived] Hernandez D, Alonso-Titos J, Vazquez T, Leon M, Caballero A, Cobo MA, Sola E, Lopez V, Ruiz-Esteban P, Cruzado JM, Sellares J, Moreso F, Manonelles A, Torio A, Cabello M, Delgado-Burgos J, Casas C, Gutierrez E, Jironda C, Kanter J, Seron D, Torres A. Clinical Relevance of Corticosteroid Withdrawal on Graft Histological Lesions in Low-Immunological-Risk Kidney Transplant Patients. J Clin Med. 2021 May 7;10(9):2005. doi: 10.3390/jcm10092005. PMID 34067039
- [Derived] Hernandez D, Vazquez T, Alonso-Titos J, Leon M, Caballero A, Cobo MA, Sola E, Lopez V, Ruiz-Esteban P, Cruzado JM, Sellares J, Moreso F, Manonelles A, Torio A, Cabello M, Delgado-Burgos J, Casas C, Gutierrez E, Jironda C, Kanter J, Seron D, Torres A. Impact of HLA Mismatching on Early Subclinical Inflammation in Low-Immunological-Risk Kidney Transplant Recipients. J Clin Med. 2021 Apr 29;10(9):1934. doi: 10.3390/jcm10091934. PMID 33947168

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 230 patients, 125 were not randomized because of: screening failure 74; patient wishes 16; acute rejection 9; graft loss 9; died 3; lost to follow-up 1 and other causes 13. The main causes of screening failure were: creatinine >2 mg/dl and subclinical rejection in the protocol biopsy at the third month. 105 patients were finally included
Period: Overall Study
Arm/Group | Steroids, Tacrolimus and Mycophenolate | Tacrolimus and Mycophenolate
Started | 52 | 53
Completed | 39 | 36
Not Completed | 13 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Steroids, Tacrolimus and Mycophenolate | Tacrolimus and Mycophenolate | Total
Number analyzed (Participants) | 52 | 53 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 44 | 87
  >=65 years | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (10) | 52.1 (14) | 53.4 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 39 | 38 | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race / Ethnicity: Caucasian | 47 | 51 | 98
  Race / Ethnicity: Black | 3 | 1 | 4
  Race / Ethnicity: North African | 1 | 1 | 2
  Race / Ethnicity: Hispanic | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Spain | 52 | 53 | 105

OUTCOME MEASURES:

1. Primary Outcome: Cases of Kidney Transplant Patients With DSA
Description: Measurements of DSA at baseline, and at 3, 6, 12, 18 and 24 months
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroids, Tacrolimus and Mycophenolate | Tacrolimus and Mycophenolate
Number analyzed (Participants) | 39 | 36
Participants | 0 | 0

2. Secondary Outcome: Mean Score on the Protocol Biopsies in the Two Treatment Groups
Description: Measurement at 24 months according to the Banff classification. The Banff Classification of Allograft Pathology is an international consensus classification for the reporting of biopsies from solid organ transplant. The scale ranges from 0 to 3, 3 being the worst.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroids, Tacrolimus and Mycophenolate | Tacrolimus and Mycophenolate
Number analyzed (Participants) | 28 | 26
score on a scale
  Interstitial fibrosis and tubular atrophy | 1.18 (1.14) | 1.83 (1.5)
  Chronic graft lesion | 1.96 (1.5) | 2.6 (1.5)
  Glomerulitis | 0.17 (0.4) | 0.08 (0.3)
  Peritubular capillaritis | 0.24 (0.6) | 0.20 (0.5)
  Tubulitis | 0.5 (0.7) | 0.56 (0.6)
  Interstitial inflammation | 0.82 (0.7) | 0.68 (0.7)
  Arteritis | 0 (0) | 0 (0)
  Interstitial fibrosis | 0.6 (0.62) | 0.88 (0.78)
  Tubular atrophy | 0.6 (0.56) | 0.88 (0.8)
  Graft glomerulopathy | 0.14 (0.45) | 0 (0)
  Chronic vascular lesions | 0.58 (0.9) | 0.64 (0.7)
  Arteriolar hyalinosis | 0.53 (0.7) | 0.69 (0.8)

3. Secondary Outcome: Number of Participants With Acute Rejection Lesions
Description: Patients with acute rejection lesions (including subclinical rejection) at 24 months according to Banff classification
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroids, Tacrolimus and Mycophenolate | Tacrolimus and Mycophenolate
Number analyzed (Participants) | 28 | 26
Participants | 2 | 3

4. Secondary Outcome: Incidence of Diabetes Mellitus
Description: Incidence of diabetes mellitus after kidney transplant in both groups at 1, 2, 3, 4, 6, 9, 12, 18 and 24 months
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroids, Tacrolimus and Mycophenolate | Tacrolimus and Mycophenolate
Number analyzed (Participants) | 39 | 36
Participants | 10 | 6

5. Secondary Outcome: Lipid Profile
Description: Lipid profile after kidney transplant in both groups at 24 months
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Steroids, Tacrolimus and Mycophenolate | Tacrolimus and Mycophenolate
Number analyzed (Participants) | 39 | 36
mg/dl
  Cholesterol | 164 (28) | 161 (27)
  HDL | 51 (14) | 44.7 (10)
  LDL | 86 (21) | 92 (18)
  Triglycerides | 140 (54) | 127 (7.8)

6. Secondary Outcome: Blood Pressure
Description: Blood pressure after kidney transplant in both groups at 24 months
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Steroids, Tacrolimus and Mycophenolate | Tacrolimus and Mycophenolate
Number analyzed (Participants) | 39 | 36
mmHg
  Systolic BP | 133 (16) | 125 (15)
  Diastolic BP | 74.9 (11) | 76 (9.7)

7. Secondary Outcome: Renal Function
Description: Renal function after kidney transplant in both groups at 24 months measured according to the creatinine (mg/dL) concentrations
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Steroids, Tacrolimus and Mycophenolate | Tacrolimus and Mycophenolate
Number analyzed (Participants) | 39 | 36
mg/dl | 1.34 (0.4) | 1.4 (0.4)

8. Secondary Outcome: Assess the Adherence to Immunosuppressive Therapy in the Two Treatment Groups
Description: The Basle scale was used to assess adherence (BAASIS questionnaire) to immunosuppressive therapy.
Time Frame: At 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroids, Tacrolimus and Mycophenolate | Tacrolimus and Mycophenolate
Number analyzed (Participants) | 39 | 36
Participants
  Forgot at least one dose during last 4 weeks | 0 | 1
  Dose taken 2 hours or more before or after time | 3 | 11

9. Secondary Outcome: Patient Survival
Description: Patient survival after kidney transplant in both groups
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroids, Tacrolimus and Mycophenolate | Tacrolimus and Mycophenolate
Number analyzed (Participants) | 39 | 36
Participants | 39 | 36

10. Secondary Outcome: Graft Survival
Description: Graft survival after kidney transplant in both groups
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroids, Tacrolimus and Mycophenolate | Tacrolimus and Mycophenolate
Number analyzed (Participants) | 39 | 36
Participants | 39 | 36

11. Secondary Outcome: Renal Function
Description: Renal function after kidney transplant in both groups at 24 months measured according to the proteinuria (mg/24 h) concentrations
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: mg/24h
Arm/Group | Steroids, Tacrolimus and Mycophenolate | Tacrolimus and Mycophenolate
Number analyzed (Participants) | 39 | 36
mg/24h | 209 (185) | 148 (82)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Steroids, Tacrolimus and Mycophenolate | Tacrolimus and Mycophenolate
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/53
Serious Adverse Events (participants affected / at risk) | 10/52 | 15/53
Other Adverse Events (participants affected / at risk) | 0/52 | 0/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Steroids, Tacrolimus and Mycophenolate (N=52) | Tacrolimus and Mycophenolate (N=53)
Infection (Renal and urinary disorders) | 5 | 12 — Infection requiring attention
Cardiovascular Disease (Cardiac disorders) | 3 | 2
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT02284464/Prot_SAP_000.pdf